CLINICAL TRIAL: NCT05460013
Title: Impact of Oral Nutritional Supplements on Nutritional, Gut Functional and Clinical Outcomes: a Randomized Controlled Trial in Patients Undergoing Haematopoietic Stem Cell Transplantation
Brief Title: Impact of Oral Nutritional Supplements on Patients Undergoing Haematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-M05
Record Dates: First submitted 2022-07-05; First posted 2022-07-15 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Haematological Malignancy
Keywords: Hematopoietic Stem Cell Transplantation; Oral Nutritional Supplements; Body Weight; Body Composition
MeSH Terms: conditions — Hematologic Neoplasms; Body Weight | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Control (Placebo Comparator)
  Interventions: Dietary Supplement: Traditional Control
- Oral Nutritional Intervention (Experimental)
  Interventions: Dietary Supplement: Oral Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Traditional Control — Placebo control is a compounded made-up shake that is traditionally used by the Haematology ward to supplement patients receiving HSCT. The control provides an equivalent of 500kcals and 20.6g protein, 3.4g fiber per day. The participants will be randomly assigned to consume the control twice daily for the duration of 7 days prior to the admission to the day of discharge.
  Arms: Placebo Control
Dietary Supplement: Oral Nutritional Supplement — The product to be studied is a standard polymeric formula. It is intended to provide 500cals, 18.4g protein, and 5g fiber per day. The fiber contained is mostly presented in the form of soluble fiber (inulin, fructo-oligosaccharide). The participants will be randomly assigned to consume the intervention twice a day for the duration of 7 days prior to the admission to the day of discharge.
  Other Names: Ensure Complete (Abbott)
  Arms: Oral Nutritional Intervention

SUMMARY:
Malnutrition is common after haematopoietic stem cell transplantation (HSCT), and is a well-known prognostic factor for survival. HSCT-associated treatments are metabolic and digestively intolerant, hence can induce a significant reduction in oral intake. Thus weight loss, as well as a reduction in serum albumin, and pre-albumin levels, are frequent following HSCT. Although the gut remains functional, sore mouth, mucositis, dysphagia, nausea, vomiting, and diarrhoea will inevitably hinder the implementation of enteral nutrition (EN), thus leading to a deficit between daily intake and requirement. Side effects of chemotherapy and antibiotics in combine will contribute to the alteration of intestinal flora on top of the existing gut symptoms, further impairing nutrient digestion and absorption.

Oral nutritional supplements (ONS) are foods for special medical purposes (FSMP) that are specially formulated for oral nutritional support. Limited retrospective studies performed in Western countries have found that ONS was tolerable for HSCT patients eligible for EN, however, the data is sparse in China to support the safety of usage amongst this population. On the other side, what is less clear is the nature of soluble fiber upon the intestinal microenvironment in patients undergoing HSCT. It would be worthwhile to investigate the impact of fibre-modulated ONS on gut function and symptoms.

The study is a prospective study. All the participants will be recruited from a single research center (Renji Hospital). The participants will be randomized into two groups: traditional treatment or ONS. Ensure complete (Abbott), which contains soluble dietary fiber such as fructo-oligosaccharide (FOS) and inulin, will be served as the ONS for testing.

The primary aim of the study is to examine the between-group change from baseline body weight at 28 days post-transplantation. The secondary outcomes include the within-group and between-group dynamic change in the peri-transplant period for the following: body weight, fat-free mass, circumference, handgrip test, and patient-generated global subjective assessment. The tolerability of supplementing ONS and its' effect on gut function as well as on infection rate is also of interest.

DETAILED DESCRIPTION:
Standard Operating Procedures:

The study is located in Renji Hospital Stem Cell Transplant Unit, including Haematology Outpatient Department and Clinical Nutrition Department. All the patients aged between 18 and 75 years planned for HSCT and who are able to understand and sign an informed consent form are eligible for the study. The potential participants will be provided with the information sheet by the dietitian on the day of their outpatient pre-assessment visit. Each participant will be allocated with a study-specific code to protect their confidentiality. After recruitment, the participants will be asked to consume either the placebo control OR the ONS for testing, intended for supplementation for the duration of 7 days prior to HSCT admission. Anthropometry, biochemistry, and functional assessments are planned at four time points: before admission (baseline), the day of transplantation (D0), 14 days post-transplantation (D14) and 28 days post-transplantation (D28). In addition, nutritional intakes and gut assessments will be collected for the duration of the whole admission. If a subject is discharged home before D14 or D28, then these will be attempted at the appropriate time when the patient attended Haematology Outpatients for medical follow-up visits. Teleconsultation might be involved if the visit is not possible. All the data will be stored in an electronic database. It will be password protected with access only restricted to major investigators. All adverse events occurring within the trial will be collected at each visit for assessment of safety.

Sample Size Assessment:

A total number of 100 participants is determined necessary to demonstrate an effect. This sample size is designed to provide 85% power to detect a 1.2kg difference in body weight using an alpha=0.05(two-sided) to account for comparisons.

Plan for missing data:

A variable could be reported as missing by reasons possibly associated with logistic issues or participants declined to take the measurements. Strategy to minimize missing data includes setting up planning and time schedule in the Excel sheet to keep all the investigators notified.

Statistical Analysis Plan:

The demographic and clinical characteristics of patients will be summarized using descriptive statistics. Data analysis will be carried out using Statistical Analysis System (SAS) 9.4. Statistical analysis software. The mean or median change in continuous variables between the group by time points is assessed using t-test or Wilcoxon's rank sum test. Changes in categorical variables is assessed using Pearson chi-square or McNemar's test. Analysis of covariance or Analysis of variance might be applied as needed.

ELIGIBILITY:
Inclusion Criteria:

* Planned for HSCT
* No contraindications to enteral nutrition
* Able to consent

Exclusion Criteria:

* Existing contraindications to enteral nutrition
* Existing infectious diarrhoea
* Had other malignancies
* Had gut surgery in a year
* Had used prebiotics or probiotics or synbiotic in a month
* Immunosuppressive OR prolonged corticosteroid therapy (more than three months)
* Chronic kidney disease (eGFR < 60 mL/min/1.73m2)
* Pregnancy or lactation
* Had an allergy, or intolerance to ingredients of dietary supplements
* Judged to be unsafe to tolerate fiber

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The between-group change for body weight | Change from baseline in body weight at 28 days post transplantation
  Body weight is assessed in kilograms

SECONDARY OUTCOMES:
The within-group change for body weight | Change from baseline in body weight at the day of transplantation, 14 days post transplantation and 28 days post transplantation
  Body weight is assessed in kilograms
The within-group and between-group change for fat free mass | Change from baseline in fat free mass at the day of transplantation, 14 days post transplantation and 28 days post transplantation
  Fat free mass is assesses in kilograms
The within-group and between-group change for calf circumference | Change from baseline in calf circumference at the day of transplantation, 14 days post transplantation and 28 days post transplantation
  Calf circumference is assessed in centimeter
The within-group and between-group change for handgrip test | Change from baseline in handgrip test at the day of transplantation, 14 days post transplantation and 28 days post transplantation
  Handgrip test is assessed in kilograms
The within-group and between-group change for Patient-Generated Subjective Global Assessment | Change from baseline in PG-SGA at 28 days post transplantation
  Patient-Generated Subjective Global Assessment (PG-SGA) is an universally used nutritional assessment tool. It is assessed in percentage based on the rated scores.
The within-group and between-group change for microbiota diversity | Change from baseline in faecal microbe diversity as well as gut microbiota-derived metabolites in urine and blood at the day of discharge
  The diversity is assessed through faecal, blood and urine sample
The within-group and between-group change for gut symptoms | Change from baseline in gut symptoms at the day of transplantation, 14 days post transplantation and 28 days post transplantation
  Gut symptoms is assessed through the presence of diarrhoea and bloating in percentage
The between-group change for infection rate | at 28 days post transplantation
  Infection rate is assessed in percentage
The tolerability of supplementing the standard polymeric formula in the targeted population | at 28 days post transplantation
  This refers to the drop-out rate

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China